CLINICAL TRIAL: NCT05644171
Title: RESTORES Trial: RESToration Of Rehabilitative Function With Epidural Spinal Stimulation
Acronym: RS-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Neuroscience Institute (Other)
Collaborators: Agency for Science, Technology and Research (Other); Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS-01
Record Dates: First submitted 2022-10-30; First posted 2022-12-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Spinal Cord Injury
Keywords: Spinal cord injury; Epidural spinal stimulation; Implantation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with motor complete chronic spinal cord injury (Other)
  Interventions: Device: RESToration Of Rehabilitative function with Epidural spinal Stimulation

INTERVENTIONS:
Device: RESToration Of Rehabilitative function with Epidural spinal Stimulation — 15 patients with chronic motor SCI will be recruited in total for this study. The recruited patients will not be randomized nor blinded due to the nature of this study. Pre-op rehabilitation session will take place over 4 weeks. 1 month post-surgical implants, patients will undergo 24 weeks of rehabilitation. The training sessions may continue to take place after the stipulated 24 weeks as long the electrode remains implanted, and the patient is available.

SUMMARY:
Spinal Cord Injury (SCI), being a devastating diagnosis, has little to no recovery which leads to a long-standing of debilitating impairment for affected patients. The NNI Neurosurgery team, together with our collaborators, are expanding our recruitment from our pilot trial named RESTORES: RESToration of Rehabilitative function with Epidural Spinal Stimulation. This study aims to investigate the feasibility of electrical stimulation via a spinal cord stimulator (SCS), which will be implanted into the study subjects, and advanced robotic neurorehabilitation to aid in improving neurological function in patients diagnosed with chronic SCI. An additional 15 patients on top of the 3 ongoing patients, male and female participants, above the age of 21 who have been diagnosed with the condition for more than a year will be recruited for this study over a 2-year period. Rehab sessions will take place pre and post-surgical implant, assessing subject improvements

DETAILED DESCRIPTION:
Motor complete SCI is defined as American Spinal Injury Association (ASIA) impairment Grade A or B, with no motor function preserved below the level of injury. This in-turn results in significant catastrophic dysfunction and disability to the individual's physical and mental health, reducing quality of life and increasing caregiver burden which translates to high socioeconomic costs. The current treatments for chronic SCI involves aggressive rehabilitation to maximize residual neurological function and devices to compensate for neurological loss. However, neurological improvement is dismal, with 94.4% of patients demonstrating no neurological improvement 5-years post-injury. Experimental and electrophysiological observations revealed that spinal hide networks have the capacity to generate basic locomotor rhythmicity without supraspinal input to the cord. SCS, consisting of a small array of electrodes surgically implanted into the epidural space stimulates afferent sensory pathways in specific patterns to drive voluntary and autonomically controlled motor responses. Activity-based training in conjunction with SCS has been shown to bolster neuroplasticity and recovery caudal to the injury site. We aim to deliver epidural spinal stimulation via an implanted SCS and together with personalized advanced neuro-rehabilitation to study the improvement of neurological function after chronic SCI.

ELIGIBILITY:
⦁ Inclusion Criteria

For inclusion in the study, the potential patient has to fulfil all of the following criteria:

1. 21 years old and older
2. Chronic (greater than one year) motor complete (AIS classification A or B) SCI
3. Spinal injury between the levels of Cervical 2 (C2) to Thoracic 12 (T12)
4. Segmental reflexes that remain functional below the level of lesion
5. Able to perform the perioperative rehabilitation program as judged by the research team

   * Exclusion Criteria

Potential patients will be excluded from the trial if they fulfil any of the following criteria:

1. Significant medical co-morbidities that would significantly increase the risk of the operation
2. Severe dysautonomia with systolic blood pressure fluctuation less than 50 or more than 200mmHg on tilt table testing
3. Painful musculoskeletal dysfunction, contractures, unhealed fractures, pressure sores, severe spasticity, and osteoporosis
4. Significant psychological issues or ongoing drug abuse
5. Pregnancy and lactating patients
6. Progressive spinal cord disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by CTCAE v5.0 | 6 months
  The adverse events in patient's with proposed surgical implantation and robotic neuro-rehabilitation during the course of study will be assessed. Particularly, during the first 6 months of the study and post implantation.

SECONDARY OUTCOMES:
Assessing the improvement in motor outcomes post surgical implantation | 2 years
  Volitional control including independent locomotion with epidural spinal stimulation and robotic neuro-rehabilitation will be assessed to check for improvement in motor functions.
  This assessment will be done during rehabilitation session where the post-surgical movement results will be compared against the pre-surgical results for better understanding and study.
Assessing autonomic function post surgical implantation | 2 years
  The improvement in hemodynamic, bowel and bladder control with epidural spinal stimulation and robotic neuro-rehabilitation will be assessed continuously post surgical implantation

CONTACTS AND LOCATIONS:
Locations (1):
- National Neuroscience Institute, Singapore, Singapore

REFERENCES:
- [Background] Kirshblum S, Millis S, McKinley W, Tulsky D. Late neurologic recovery after traumatic spinal cord injury. Arch Phys Med Rehabil. 2004 Nov;85(11):1811-7. doi: 10.1016/j.apmr.2004.03.015. PMID 15520976
- [Background] Minassian K, Jilge B, Rattay F, Pinter MM, Binder H, Gerstenbrand F, Dimitrijevic MR. Stepping-like movements in humans with complete spinal cord injury induced by epidural stimulation of the lumbar cord: electromyographic study of compound muscle action potentials. Spinal Cord. 2004 Jul;42(7):401-16. doi: 10.1038/sj.sc.3101615. PMID 15124000
- [Background] Lim PA, Tow AM. Recovery and regeneration after spinal cord injury: a review and summary of recent literature. Ann Acad Med Singap. 2007 Jan;36(1):49-57. PMID 17285186
- [Background] Minassian K, Persy I, Rattay F, Pinter MM, Kern H, Dimitrijevic MR. Human lumbar cord circuitries can be activated by extrinsic tonic input to generate locomotor-like activity. Hum Mov Sci. 2007 Apr;26(2):275-95. doi: 10.1016/j.humov.2007.01.005. Epub 2007 Mar 6. PMID 17343947
- [Background] Teo SH, Sew S, Backman C, Forwell S, Lee WK, Chan PL, Dean E. Health of people with spinal cord injury in Singapore: implications for rehabilitation planning and implementation. Disabil Rehabil. 2011;33(15-16):1460-74. doi: 10.3109/09638288.2010.533812. Epub 2010 Nov 20. PMID 21091048
- [Derived] Wee SK, Valerie ZYN, Phua MW, Lui WL, Misbaah F, Ker RXJ, Ng WH, Rui Wan K. Synergistic integration of epidural spinal cord stimulation with robotic therapy and neurorehabilitation to facilitate functional recovery in chronic sensorimotor complete spinal cord injury: A case series. Adv Rehabil Sci Pract. 2025 Jun 24;14:27536351251343738. doi: 10.1177/27536351251343738. eCollection 2025 Jan-Dec. PMID 40568376
- See also: Recruitment Challenges in Spinal Cord Stimulation Trial for Motor Recovery in Patients with Chronic Complete Spinal Cord Injury — https://pubmed.ncbi.nlm.nih.gov/40507687/
- See also: Synergistic integration of epidural spinal cord stimulation with robotic therapy and neurorehabilitation to facilitate functional recovery in chronic sensorimotor complete spinal cord injury: A case series — https://pubmed.ncbi.nlm.nih.gov/40568376/